CLINICAL TRIAL: NCT03247725
Title: Pain Monitor: a Randomized Controlled Trial to Test the Efficacy of a Pain App in the Treatment of Chronic Pain
Brief Title: Efficacy of Pain Monitor, a Smartphone App for Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Principal Investigator, Carlos Suso Ribera, Principal Investigator, Universitat Jaume I
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UJI_PainMonitor
Record Dates: First submitted 2017-07-25; First posted 2017-08-14 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Three conditions. Patients will be randomly assigned to one of the three conditions.
Masking Description: Patients will be informed of the condition they have been assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment as usual (waiting list) (Active Comparator): Patients at this condition will receive the usual medical treatment at the pain unit, but they will not be monitored daily using the app.
  Interventions: Other: Treatment as usual (medical)
- Treatment as usual + app (without alarm) (Experimental): Participants at this condition will receive the usual medical treatment for their pain but also they will be monitored daily using the Pain Monitor app. Because alarms will not be generated, physicians will not know if an undesired event is occuring despite the app is actually collecting data.
  Interventions: Other: pain app; Other: Treatment as usual (medical)
- Treatment as usual + app (with alarm) (Experimental): Participants at this condition will receive the usual medical treatment for their pain but also they will be monitored daily using the Pain Monitor app. Alarms will be generated in the face of certain preestablished events. Physicians will be asked to call patients and change/stop treatment if an alarm is received.
  Interventions: Other: pain app; Other: Treatment as usual (medical)

INTERVENTIONS:
Other: pain app — Pain Monitor app has been developed by a multidisciplinary pain expert panel, including physicians, psychologists, and nurses. Content has been validated in a previous study and usability has been shown to be excellent.
  Arms: Treatment as usual + app (with alarm); Treatment as usual + app (without alarm)
Other: Treatment as usual (medical) — Patients will be offered the usual treatment for their pain, which is not changed by study participation

SUMMARY:
The present investigation aims at exploring the effect of including a pain app called Pain Monitor for chronic pain patients' daily monitoring. Three conditions will be set:

1. usual treatment (waiting list)
2. usual treatment + app (without alarms)
3. usual treatment + app (with alarms)

DETAILED DESCRIPTION:
Chronic pain is defined as one that lasts for at least three to six months, provided that this time is greater than the normal healing period of an injury. This pathology has become an important public health problem due to its high prevalence. In particular, it is estimated that it affects 20-30% of the adult population around the world. Medical interventions are the first-line treatment in recent clinical practice guidelines. Unfortunately, the effectiveness of medical interventions is only modest. Treatments significantly reduce pain on average, but the effect tends to be small . In addition, the drugs are not effective for a large percentage of patients.

What these and other research suggest is that focusing only on large sample studies and the use of average change scores calls into question the usefulness of current patient-centered treatments. As noted by Dr. Turk, when data are averaged, various pain syndromes, drugs, surgical procedures, and studies in different countries are often included, which may mask the efficacy results of different treatments with Different samples. Single case methodology could be one of the ways to overcome these limitations. The single case investigation is a type of experimental study that offers experimental control within a single case.

Some studies have already demonstrated the usefulness of these designs in chronic pain. In fact, the benefits of using this methodology as opposed to large sample studies were discussed recently during the 10th Congress of the European Pain Federation. These benefits include the need for a reduced number of participants, the ability to follow clinical evolution in real time and continuously, the amount of data provided, and applicability when using a control group is impractical or unethical.

The investigators conducting the present investigation recently conducted a study at the Pain Unit of the Vall d'Hebron Hospital to explore the effectiveness of current medical treatments. According to previous investigations, the treatment effect was only small (d = 0.32) and only a percentage of the patients (18.1%) had a clinically significant reduction of pain (ie a reduction greater than 30% ).

From these results and the literature reviewed, a single case design could be an alternative method for research in the Pain Unit. However, the implementation of this type of methodology can be very costly due to the continuous evaluation of the evolution of the patient. In this sense, several studies have already shown that mobile applications (app) can effectively control the evolution of a wide range of pathologies in health settings . In fact, a recent controlled clinical study found that ecological records performed with mobile app had greater reliability than paper-and-pencil records.

Rosser and Eccleston conducted a comprehensive review of existing apps for pain and the conclusion was that there was little evidence to support the use of current apps. Specifically, these authors showed that most apps did not specify whether their content was validated, did not include psychological components and none had been applied in a clinical study. In light of these results, Dr. Carlos Suso Ribera and Dr. Ribera Canudas contacted the research team Labpsitec of Jaume I University, who were developing an application for pain called "Pain Monitor". Dr. Carlos Suso Ribera and Dr. Ribera Canudas of the Pain Unit collaborated with Dr. Azucena García Palacios and Dr. Diana Castilla López of the Universitat Jaume I in the final development of the application of pain, Following the guidelines of Rosser and Eccleston.

App content validity and usability was tested in a previous study at the pain unit of the Vall d'Hebron Hospital (Suso-Ribera et al., in preparation). Thus, the study objective is to test if the introduction of this tool in the day-to-day work of the pain unit improves pain management of chronic pain patients. To do this, it is necessary to compare the evolution of patients who follow the usual treatment at the pain unit (without app) with a group of patients who do use the Pain Monitor app. In addition, the present study investigators have created a new utility that allows alarms to be generated by healthcare professionals in the presence of an undesired event, such as an adverse effect of the medication or a lack of response to medical treatment. Before determining that both the use of the app and this new utility (alarms) are beneficial for patient care, it is necessary to perform a clinical trial comparing the 3 conditions mentioned above:

1. usual treatment (waiting list)
2. usual treatment + app (without alarms)
3. usual treatment + app (with alarms) Therefore, this is a clinical trial without drugs. This is not an observational study since the physicians of patients in the app + alarms condition will be asked to react to an alarm (i.e., if the patient has nausea for 3 consecutive days) by calling the patient and changing the treatment telematically, if necessary, so that the patient can collect the prescription at his primary care center.

If the condition app with alarms results in a better treatment of chronic pain patients, participants of the other two conditions will be offered the possibility to use the app with alarms at the end of the study.

The study will be conducted at the Pain Unit of the Vall d'Hebron Hospital. All study procedures have been approved by the ethical committee of the Vall d'Hebron Hospital.

ELIGIBILITY:
Inclusion Criteria:

* The patient is over 18 years of age
* The patient has a mobile phone with Android operating system
* The patient has the physical ability to use the application
* The patient does not present psychological and / or cognitive alterations or problems with language that make their participation difficult
* The patient voluntarily wants to participate and signs the informed consent

Exclusion Criteria:

* The patient is under 18 years
* The patient does not have a mobile phone or has a mobile phone in which Android is not the operating system (the app is currently only available for Android for economic reasons)
* The patient does not have the physical capacity to use the application
* The patient does not have the capacity to participate due to psychological and / or cognitive alterations or problems with language
* The patient does not want to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity | Dialy during 30 days (app condition) in the app condition (with and without alarm)
  A numerical rating scale (0-10 range) will be used.
Change in side effects | Dialy during 30 days (app condition) in the app condition (with and without alarm)
  A list of the most frequent side effects of pain medication was created
Change in pain intensity | Twice (first day of study and 30 days after, at the end of study) in the TAU condition
  A numerical rating scale (0-10 range) will be used.
Change in side effects | Twice (first day of study and 30 days after, at the end of study) in the TAU condition
  A list of the most frequent side effects of pain medication was created

SECONDARY OUTCOMES:
Change in mood | Dialy during 30 days (app condition) in the app condition (with and without alarm)
  Questionnaire on mood validated against the Profile of Mood States
Change in mood | Twice (first day of study and 30 days after, at the end of study) in the TAU condition
  Questionnaire on mood validated against the Profile of Mood States
Change in rescue medication use | Dialy during 30 days (app condition) in the app condition (with and without alarm)
  Amount of rescue medication will be assessed
Change in rescue medication use | Twice (first day of study and 30 days after, at the end of study) in the TAU condition
  Amount of rescue medication will be assessed
Change in pain interference | Dialy during 30 days (app condition) in the app condition (with and without alarm)
  Interference of pain with patient's life
Change in pain interference | Twice (first day of study and 30 days after, at the end of study) in the TAU condition
  Interference of pain with patient's life
Change in general health | Dialy during 30 days (app condition) in the app condition (with and without alarm)
  A general health item was validated against the phsyical health scale of the Short Form 12
Change in general health | Twice (first day of study and 30 days after, at the end of study) in the TAU condition
  A general health item was validated against the phsyical health scale of the Short Form 12
Change in fear of pain | Dialy during 30 days (app condition) in the app condition (with and without alarm)
  2 items validated against the Fear Avoidance Beliefs Scale
Change in fear of pain | Twice (first day of study and 30 days after, at the end of study) in the TAU condition
  2 items validated against the Fear Avoidance Beliefs Scale
Change in pain acceptance | Dialy during 30 days (app condition) in the app condition (with and without alarm)
  2 items validated against the Chronic Pain Acceptance Questionnaire
Change in pain acceptance | Twice (first day of study and 30 days after, at the end of study) in the TAU condition
  2 items validated against the Chronic Pain Acceptance Questionnaire
Change in pain catastrophizing | Dialy during 30 days (app condition) in the app condition (with and without alarm)
  3 items validated against the Pain Catastrophizing Scale
Change in pain catastrophizing | Twice (first day of study and 30 days after, at the end of study) in the TAU condition
  3 items validated against the Pain Catastrophizing Scale

CONTACTS AND LOCATIONS:
Overall Officials: Ángela Mesas Idáñez, MD, Principal Investigator — Staff Doctor
Locations (1):
- Vall d'Hebron Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Only the two principal investigators, Dr. Mesas and Dr. Suso, will be able to access to individual participant data.

REFERENCES:
- [Background] Rosser BA, Eccleston C. Smartphone applications for pain management. J Telemed Telecare. 2011;17(6):308-12. doi: 10.1258/jtt.2011.101102. Epub 2011 Aug 15. PMID 21844177
- [Derived] Suso-Ribera C, Mesas A, Medel J, Server A, Marquez E, Castilla D, Zaragoza I, Garcia-Palacios A. Improving pain treatment with a smartphone app: study protocol for a randomized controlled trial. Trials. 2018 Feb 27;19(1):145. doi: 10.1186/s13063-018-2539-1. PMID 29482614